CLINICAL TRIAL: NCT00506194
Title: Short-Term Intensive Insulin Therapy Induction of Long-term Glycemic Control Is Associated With Improvement of ß-Cell Function in Newly Diagnosed Type 2 Diabetic Patients
Brief Title: Short-Term Intensive Insulin Therapy Induction of Long-term Glycemic Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGH 94-09-09
Record Dates: First submitted 2007-07-24; First posted 2007-07-25 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; oral glucose tolerance test; insulin; oral anti-diabetic drug; ß-cell function
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Insulin; Isophane Insulin, Human; Insulin Glargine; Metformin; glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin (Experimental): Insulin therapy was initiated at a 75% total daily dose in the last day hospitalization with Insulatard. Two third of daily dose was administered before breakfast and the other was administered at bedtime. Insulin doses were titrated every 3 days to achieve target FPG and pre-supper blood glucose values between 90 and 130 mg/dl. Bedtime insulin doses were titrated based on FPG values and the pre-breakfast dose was titrated base on pre-supper blood glucose.
  Interventions: Drug: Insulin
- OAD (Active Comparator): Subject in other OAD group was visited every two weeks in the two months and the every four weeks. The subjects will start with Gliclazide-MR 30mg before breakfast, The dosage was titrated based on the fasting blood glucose on the visiting day with the same target. Decreased by 30mg if blood glucose was <70mg /dl, decreased by 15 mg if blood glucose was 70-90mg/dl, no change if blood glucose was 90-130mg/dl, increased by 15 mg if blood glucose was 131-160 mg/dl, increased by 30 mg if blood glucose >160mg/dl. When the Gliclazide-MR dose each to the maximum dose of 60 mg twice daily, Metformin was added. The titration of Metformin was use 250mg for an adjust dosage with the same target.
  Interventions: Drug: OAD

INTERVENTIONS:
Drug: Insulin
  Other Names: Insulatard, Actrapid, Lantus, monotard
  Arms: Insulin
Drug: OAD — Gliclazide-MR, Metformin, Glimepiride
  Other Names: Diamicron-MR, Glucophage, Amaryl
  Arms: OAD

SUMMARY:
We designed this prospective, randomized control study to compare the benefits between the insulin therapy and OADs after correction of the glucose toxicity with a short period of intensive insulin therapy.

DETAILED DESCRIPTION:
OBJECTIVE-Type 2 diabetes is associated with defects in insulin secretion and insulin action. Hyperglycemia may aggravate these defects, a feature known as glucose toxicity. Previous studies have shown that acute correction of hyperglycemia in subjects with long-standing type 2 diabetes gives only short-term improvement in glycemic control after discontinuation of insulin. The current study attempts to identify any characteristics of patients with newly diagnosed type 2 diabetes (fasting glucose >300mg/dL) who would have a long-term benefit, in terms of glycemic control, from a brief course of insulin therapy.

RESEARCH DESIGN AND METHODS-Newly diagnosed type 2 diabetic patients with severe hyperglycemia (fasting blood glucose >300 mg/dL or random blood glucose >400 mg/dL) will be hospitalized and treated with intensive insulin injection for 10 to 14 days. Oral glucose tolerance will be performed after one week of intensive insulin treatment. After discharge, patients will be randomized to receive insulin injection or oral anti-diabetic drug for further management. Patients will be followed in our clinics and adjust their medication according to their blood glucose levels. Oral glucose tolerance test will be repeated 6 months later, whereas the insulin sensitivity and beta-cell function will be evaluated again.

EXPECTED RESULTS-We will respect that short-term intensive insulin therapy can induce lone-term glycemic control in newly diagnosed type 2 diabetes with severe hyperglycemia.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed type 2 diabetic patients.
2. Hospitalization due to hyperglycemia hyperosmolality syndrome.
3. Those who age between 30 and 80 years old and can inject insulin by themselves.

Exclusion Criteria:

1. Pregnant women.
2. Impaired liver function (ALT > 120 U/L)
3. Impaired renal function (Serum creatinine >3.0 mg/dL)
4. Recently suffered from MI or CVA.
5. Patients are acute intercurrent illness.
6. 2-hour C-peptide level < 1.8 ng/mL.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2005-10; Primary Completion 2007-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Short-term intensive insulin therapy can decrease the insulin resistance and improve the Beta-cell function in newly diagnosed type 2 diabetes with severe hyperglycemia. | 6 months

SECONDARY OUTCOMES:
Improve long term glycemic control | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Harn-Shen Chen, MD, PhD, Principal Investigator — Division of endocrinology and metabolism, Department of medicien, Taipei Veterans General Hospital
Locations (1):
- Division of Endocrinology and Metabolism, Department of Medicine, Taipei, Taiwan

REFERENCES:
- [Derived] Chen HS, Wu TE, Jap TS, Hsiao LC, Lee SH, Lin HD. Beneficial effects of insulin on glycemic control and beta-cell function in newly diagnosed type 2 diabetes with severe hyperglycemia after short-term intensive insulin therapy. Diabetes Care. 2008 Oct;31(10):1927-32. doi: 10.2337/dc08-0075. Epub 2008 Jun 12. PMID 18556343